CLINICAL TRIAL: NCT00496613
Title: Chemotherapy-Induced Cognitive Change and DNA Damage in Breast Cancer Survivors
Brief Title: Chemotherapy-Induced Changes to Cognition and DNA in Breast Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 07-090
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer; Long-Term Survivors
Keywords: Breast cancer; survivor
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- 1: Breast cancer survivors (2-6 years post-treatment) who were post-menopausal at the time of diagnosis and treated with a combination of chemotherapy and hormonal therapy, matched on age and education
  Interventions: Behavioral: Mini-Mental State Exam and Blood draw
- 2: Breast cancer survivors (2-6 years post-treatment) who were post-menopausal at the time of diagnosis and treated with hormonal therapy only matched on age and education
  Interventions: Behavioral: Mini-Mental State Exam and Blood Draw
- 3: Healthy women matched on age and education
  Interventions: Behavioral: Mini-Mental State Exam and Blood Draw

INTERVENTIONS:
Behavioral: Mini-Mental State Exam and Blood draw — The neuropsychological testing will be conducted by a psychometrician who will be trained and supervised by Dr. Correa. It should take approximately 2 hours to complete.Two blood samples will be collected in green top tubes for analysis of DNA damage
  Groups: 1
Behavioral: Mini-Mental State Exam and Blood Draw — The neuropsychological testing will be conducted by a psychometrician who will be trained and supervised by Dr. Correa. It should take approximately 2 hours to complete.Two blood samples will be collected in green top tubes for analysis of DNA damage
  Groups: 2
Behavioral: Mini-Mental State Exam and Blood Draw — The neuropsychological testing will be conducted by a psychometrician who will be trained and supervised by Dr. Correa. It should take approximately 2 hours to complete.Two blood samples will be collected in green top tubes for analysis of DNA damage
  Groups: 3

SUMMARY:
The purpose of this study is to learn more about how chemotherapy affects an individual's thinking abilities (cognition). Some research has shown that chemotherapy can cause changes in cognition in breast cancer survivors. However, it is not clear why this change occurs. In this study, the investigators will look to see if damage to DNA is related to these changes in cognition. Specifically, the investigators want to see 1) if women who have been treated with chemotherapy have more DNA damage than healthy women; and 2) if DNA damage is related to cognitive problems in breast cancer survivors and healthy women.

DETAILED DESCRIPTION:
The primary objective of this proposal is to obtain preliminary data regarding the association between DNA damage and cognitive functioning in breast cancer survivors. Specifically, we predict that:

1. Breast cancer survivors treated with chemotherapy and hormonal therapy will have higher levels of DNA damage as measured by the Comet assay as compared to age and education matched survivors treated with hormonal therapy only and healthy controls.
2. Survivors who meet criteria for cognitive impairment will have higher levels of DNA damage as compared to cancer survivors who do not meet criteria for cognitive impairment and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer survivors (Stage I-III) 2-6 years post all cancer treatments, but currently receiving hormone therapy.
* History of treatment with chemotherapy and/or hormonal therapy, or hormone therapy only.
* No evidence of active/recurrent disease.
* Less than 70 years old at time of recruitment.
* Post-menopausal prior to initial treatment.
* In the judgment of the consenting professional, is able to provide informed consent.
* Patient is able to understand English, through verbal and written communication.

Exclusion Criteria:

* Recurrence of breast cancer or diagnosis of another cancer except basal cell carcinoma.
* Exposure to chemotherapy or radiation therapy for any medical condition unrelated to breast cancer.
* Neurobehavioral risk factors including history of neurological disorder, or moderate to severe head trauma (loss of consciousness > 60 min or evidence of structural brain changes on imaging).
* Neurodegenerative disorders such as Alzheimer's disease, Parkinson's disease, multiple sclerosis, etc.
* Self-reported sleep disorders that could influence cognitive functioning including sleep apnea and chronic fatigue syndrome.
* Self-reported Axis I psychiatric disorder (DSM-IV), major affective disorder (untreated), bipolar disorder, schizophrenia.
* Disorder (DSM-IV), major affective disorder (untreated), bipolar disorder, schizophrenia.
* Male.

Healthy Control Inclusion Criteria:

* Have had no diagnosis of cancer except basal cell carcinoma.
* Less than 70 years old at time of recruitment.
* Post-menopausal.
* In the judgment of the consenting professional, is able to provide informed consent.
* Patient is able to understand English, through verbal and written communication

Healthy Control Exclusion Criteria:

* Exposure to chemotherapy or radiation therapy for any medical condition.
* Neurobehavioral risk factors including history of neurological disorder, or moderate to severe head trauma (loss of consciousness > 60 min or evidence of structural brain changes on imaging).
* Neurodegenerative disorders such as Alzheimer's disease, Parkinson's disease, multiple sclerosis etc.
* Self-reported sleep disorders that could influence cognitive functioning including sleep apnea and chronic fatigue syndrome.
* Self-reported Axis I psychiatric disorder (DSM-IV), major affective disorder (untreated), bipolar disorder, schizophrenia.
* Male.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Survivors Healthy women
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-06; Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
The primary goal of this preliminary study is to examine the relationship between DNA damage and chemotherapy-induced cognitive changes in breast cancer survivors. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tim Ahles, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org